CLINICAL TRIAL: NCT03130491
Title: European Study Evaluating the EMBLOK Cerebral Embolic Protection System During Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: European Study Evaluating the EMBLOK Embolic Protection System During TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emblok, Inc. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLP002-2016
Record Dates: First submitted 2017-04-11; First posted 2017-04-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-09

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR + Embolic protection (Other): subjects with severe native aortic valve stenosis who meet the commercially approved indications for transcatheter aortic valve replacement
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR); Device: EMBLOK filter

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement (TAVR) — placement of a filter to capture and remove embolic material from entering the cerebral vascular circulation during aortic valve replacement
Device: EMBLOK filter — Embolic Filter Protection System During TAVR

SUMMARY:
The primary objective is to evaluate the performance and the treatment effect of the use of the Emblok embolic protection system use during transcatheter aortic valve replacement with respect to procedure-related cerebral embolic burden as determined by DW-MRI.

DETAILED DESCRIPTION:
The enrollment of up to thirty subjects with severe native aortic valve stenosis who meet clinically approved indications for transcatheter aortic valve replacement. The primary objective evaluates performance and treatment effect of the use of the EMBLOK. A secondary objective of this study is to analyze the safety profile and the type of captured debris from the Emblok filter after TAVR. Due to the small sample size, the study is not powered to detect a reduction in actual stroke rates. However, the potential risk of stroke will be assessed based on neurological evaluations pre and post procedure. In addition, silent ischemic damage and cerebral embolic burden will be assessed using DW MRI studies.

ELIGIBILITY:
Inclusion Criteria: Subject is between 18 and 90 years of age.Subject is scheduled to undergo transcatheter aortic valve replacement (TAVR) procedure on a native aortic valve and is qualified based on pre-operative trans-thoracic echocardiogram (TTE). Subject anatomy is compatible with correct device positioning with: Iliofemoral access compatible with a 12 French arterial access system for the EMBLOK catheter (> 4 mm vessel diameter). Ascending aorta length greater than or equal to 9 cm. Ascending aorta/aortic arch diameter less than or equal to 35mm.

Female subjects of child bearing potential must have a negative pregnancy test within 48 hours prior to the index study procedure.Subject agrees to comply with all study required visits. Subject or subject's legal representative completes written Informed Consent.

Exclusion Criteria: Subject requires an emergent procedure. Contraindications to MRI including: Subjects with any non-MRI compatible implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVI procedure, claustrophobia, planned implantation of non-MRI compatible pacemaker or implantable cardioverter defibrillator within 30 days after TAVR.

Subject has experienced a myocardial infarction within 30 days of the planned index procedure.

Subject has renal insufficiency, defined as a creatinine level > 2.5 mg/dl at the time of treatment.

Subject has documented history of stroke or TIA within prior 3 months. Subject has an ejection fraction of 30% or less. Subject has a history of intolerance, allergic reaction or contraindication to any of the study medications, including heparin, aspirin, clopidogrel or a sensitivity to contrast media or anesthesia which cannot be adequately pre-treated.

Subject has known allergy to any materials used in the EMBLOK device or allergy to intravascular contrast agents that cannot be pre-medicated.

Subject has active endocarditis or an ongoing systemic infection defined as fever within temperature > 38° C and/ or WBC > 15,000 IU.

Subjects undergoing therapeutic thrombolysis. Subject has history of bleeding diathesis or a major coagulopathy. Subject is known or suspected to be pregnant, or is lactating. Subject is currently participating in another drug or device clinical study, or has other medical illnesses that may cause the subject to be non-compliant with the protocol or confound the data interpretation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Performance Endpoint | Day 1 to post procedure
  successful insertion, placement and removal of the EMBLOK system

SECONDARY OUTCOMES:
Safety Endpoint (Rate of MACCE) | 30 days
  Rate of MACCE

OTHER OUTCOMES:
Efficacy Endpoint | 2-5 days
  Reduction in embolic burden as measured by DW-MRI at baseline compared to post procedure 2-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Azeem Latib, MD, Principal Investigator — Hospital San Raffaele
Locations (2):
- Italy (2):
  - Hospital San Donato, Milan, Milano
  - Hospital San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latib A, Mangieri A, Vezzulli P, Spagnolo P, Sardanelli F, Fellegara G, Pagnesi M, Giannini F, Falini A, Gorla R, Montorfano M, Bedogni F, Colombo A, Popma J, Merhi WM, De Marco F. First-in-Man Study Evaluating the Emblok Embolic Protection System During Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Apr 13;13(7):860-868. doi: 10.1016/j.jcin.2019.11.017. PMID 32273098